CLINICAL TRIAL: NCT04128540
Title: Analgesic Efficacy of Ultrasound Guided Erector Spinae Plane Block Versus Fentanyl Infusion in Pediatric Patients Undergoing Aortic Coarcitectomy. a Randomized Controlled Study.
Brief Title: Erector Spinae Plane Block Versus Fentanyl Infusion in Pediatric Patients Undergoing Aortic Coarcitectomy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Mina Kamal Harees Abdo, Assistant Lecturer, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MD-213-2019
Record Dates: First submitted 2019-10-15; First posted 2019-10-16 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Aortic Coarctation; Erector Spinae Plane Block; Paediatric
MeSH Terms: conditions — Aortic Coarctation | interventions — Fentanyl

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control group (Other): This group will receive fentanyl infusion only
  Interventions: Drug: Fentanyl
- ESPB group (Active Comparator): This group will receive fentanyl infusion plus Ultrasound guided ESPB
  Interventions: Drug: Fentanyl; Procedure: Erector spinae plane block

INTERVENTIONS:
Drug: Fentanyl — fentanyl infusion at a dose of (1 μg/kg/hour) after induction of anesthesia and to be continued all through the whole operation.rescue analgesia by a bolus of (Fentanyl 1mcg/kg) will be given to the patients in either group, if either systolic blood pressure or heart rate increased more than 20% of the baseline readings.
Procedure: Erector spinae plane block — ultrasound guided erector spinae plane block by injecting 0.4ml/kg (1:1 solution of bupivacaine 0.25% and lidocaine 1%). This will be performed at the same side of the planned thoracotomy under strict aseptic precautions.A high frequency 12 MHz linear ultrasound transducer will be placed in a longitudinal orientation 3 cm lateral to the T3 spinous process corresponding to the T2 transverse process.
  Three muscles; trapezius, rhomboids major, and erector spinae will be identified superior to the hyperechoic transverse process.
  Using in-plane approach a 25 G needle will be inserted in caudal-cephalic direction, until the tip is deep to erector spinae muscle.
  Correct needle tip location will be confirmed by injecting 3 mL of normal saline and visualizing the linear LA spread in the fascial plane between the erector spinae muscle and the transverse process..
  Arms: ESPB group

SUMMARY:
Pain is considered to be subjective, however in children it is believed to be felt rather than expressed, because they often depend on the caregiver for their safety and well-being.

There is significant pain after thoracotomy surgery because of pleural and muscular damage, ribcage disruption, and intercostal nerve damage during surgery, which if not effectively managed, it will lead to various systemic complications; pulmonary (atelectasis, pneumonia, and stasis of bronchial secretions), cardiovascular (increased oxygen consumption and tachycardia), musculoskeletal (muscle weakness), increased neuro-hormonal response and prolonged hospital stay. So adequate and sufficient post-operative analgesia for paediatric patients is mandatory.

The use of highly potent opioids for paediatric cardiac anaesthesia has gained widespread popularity during the last 20 years.In addition to the important advantage of hemodynamic stability, the large-dose opioid-based anaesthetic techniques also blunt the stress response, However, large doses can cause oversedation, respiratory depression, and prolonged mechanical ventilation after surgery.

Erector Spinae Plane Block (ESPB), recently developed by Forero et al, is a novel technique in management of thoracic neuropathic pain guided by ultrasound. It became popular because it is much safer and easily administered than other alternative regional techniques as thoracic paravertebral and thoracic epidural block.

To our knowledge, Erector Spinae Plane Block (ESPB) performed in aortic coarcitectomy operations has not been investigated yet.This has encouraged the performance of the present study.

DETAILED DESCRIPTION:
Our study will be designed to estimate and compare the analgesic effect of single shot erector spinae plane block in pediatric patients undergoing aortic coarcitectomy via thoracotomy incision versus fentanyl infusion as the control group. Our primary outcome will be the total dose of intraoperative fentanyl bouluses.

Randomization will be achieved by using an online random number generator. Patient codes will be placed into sequentially numbered sealed opaque envelopes by a research assistant who is not involved in the study. A medical personnel not involved in patient management will be responsible for opening the envelope and give the instructions contained within each envelope to the anesthesiologist who is expert in doing the ESPB in patients included within the block group. this expert anaesthesiologist will not be involved in collecting data but another anaesthesia doctor will be responsible for patient management and collecting the intraoperative and postoperative data.

The study will be conducted in the pediatric cardiothoracic operation theatre in Abu El Reesh Pediatric Hospital -Cairo University on 28 pediatric patients aged 3 months-12 months, ASA III undergoing aortic coarcitectomy (with thoracotomy incision).

All patients will attend at the pre- anesthesia room with their parents 1 hour before the procedure after taking approval of research ethical comittee and informed consent.

Detailed history from the parents will be taken followed by a full and detailed clinical examination of the child then all investigations including CBC, coagulation profile, liver enzymes, kidney function tests, Chest x-ray ,echocardiography and blood grouping will be checked.

ECG, pulse oximetry and non-invasive blood pressure will be applied to all patients. All patients will be premedicated by intramuscular midazolam 2mg/Kg and atropine 0.2 mg/Kg 20 minutes before induction of anesthesia.

Anesthesia will be induced in all patients by sevoflurane 5% in 100% O2 followed by Placement of peripheral I.V cannula and IV administration of fentanyl (1-2µg/kg). Oral endotracheal intubation will be facilitated by IV atracurium 0.5 mg/kg and then capnogram will be connected to monitor End-tidal CO2 and muscle relaxation will be maintained by atracurium infusion in a dose of 0.5 mg/ kg/ hr.

All patients will be mechanically ventilated using pressure controlled mode with FiO2 50%, positive end expiratory pressure (PEEP) 5 cmH2O,I: E ratio of 1:2,peak inspiratory pressure (PIP) will be set to deliver a tidal volume of 6-8 ml/kg and respiratory rate will be 15 to 35 cycle / minute according to the age. our aim is to keep end tidal CO2 between 30-40 mmHg.

Sevoflurane will be used for maintenance of anaesthesia and its MAC will be determined by using bispectoral index (targeting 40-60) to standardize the depth of anaesthesia.

After insertion of a central venous catheter and an arterial cannula , nasopharyngeal temperature probe will be placed and the patient's position will be changed from supine to right lateral position.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 3 months-12 months.
2. A III .
3. Patients undergoing aortic coarcitectomy operation undergone with Lateral thoracotomy incision.

Exclusion Criteria:

1. Patients whose parents or legal guardians refusing to participate.
2. Preoperative mechanical ventilation.
3. Preoperative inotropic drug infusion.
4. Patients undergoing aortic coarctectomy operation undergone with midline sternotomy incision.
5. Known or suspected coagulopathy.
6. Any congenital anomalies of the sacrum/the vertebral column or any infection at the site of injection.
7. Known or suspected allergy to any of the studied drugs.
8. Elevated liver enzymesmore than the normal values.
9. Renal function impairment (Creatinine value more than 1.2mg/dl or blood urea nitrogen more than 20mg/dl).

Ages: 3 Months to 12 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-07-30 (Actual)

PRIMARY OUTCOMES:
The total dose of intraoperative fentanyl boluses. | From skin incision till 5 minutes after skin closure
  microgram/kg

SECONDARY OUTCOMES:
Face, Leg, Activity, Cry, Consolability | 30 min, 60 min, 2 hours, 4hours, 8hours, 16hours and 24 hours postoperatively
  1. Face
     * 0: if patient has a relaxed face
     * 1: if patient has a worried look ,eyes partially closed, mouth pursed
     * 2: if patient has deep furrows in the forehead, with closed eyes, open mouth.
  2. Legs
     * 0: if patient has usual tone and motion to limbs.
     * 1: if patient has increase tone, rigidity.
     * 2: if patient has hyper tonicity, legs pulled tight, exaggerated flexion/extension of limbs.
  3. Activity
     * 0: if patient moves easily and freely.
     * 1: if patient shifts positions, guarding.
     * 2:if patient is in fixed position, side-to-side head movement.
  4. Cry
     * 0: if patient has no cry/moan awake or asleep
     * 1: if patient has occasional moans, cries.
     * 2: if patient has frequent/continuous moans, cries, grunts.
  5. Consolability
     * 0: if patient is calm and does not require consoling
     * 1: if patient responds to comfort by touch or talk in ½- 1 minute
     * 2: if patient requires constant comforting or unable to console.
postoperative Morphine | 30 minutes postoperative till 24 hours postoperative
  mg/kg

CONTACTS AND LOCATIONS:
Locations (1):
- Kasr Al-Ainy Hospital, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided